CLINICAL TRIAL: NCT05317780
Title: Expanded Access Trial of Systemic Delivery of Aspartoacylase ASPA (rAAV9-CB6-AspA) Gene Vector in a Single Patient With Canavan Disease
Brief Title: Canavan-Single Patient IND
Status: No longer available | Type: Expanded Access
Sponsor: University of Florida (Other)
Collaborators: University of Miami (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Other Study IDs: 201601620
Record Dates: First submitted 2022-03-24; First posted 2022-04-08 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Canavan Disease
Keywords: Gene Therapy
MeSH Terms: conditions — Canavan Disease

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: rAAV9-CB6-AspA — This study is an open label, expanded access trial of a simultaneous, single intravenous (IV) and intracerebroventricular (ICV) administration of rAAV9-CB6-AspA in a child with Canavan disease. The subject will also receive an immunosuppression protocol to prevent reaction to ASPA and vector capsids.

SUMMARY:
A recombinant virus vector constructed from adeno-associated virus (AAV) has been engineered to carry the human aspartoacylase (ASPA) gene expressed from a modified CMV-enhancer chicken β-actin (CB6) promoter. The construct has been shown to produce ASPA in animal models of Canavan disease, which closely match the proposed human study. The proposed clinical trial is an open label, expanded access study administering rAAV9-CB6-AspA gene vector by simultaneous systemic and intracerebroventricular routes to a single human subject (18-24 months of age) with Canavan disease. The subject will also receive immune modulation to transiently ablate B-cells (Rituximab) and modulate T-cell response (Sirolimus) prior to the initial exposure to AAV9. Given the null AspA mutations of the subject and current AAV seronegative status, this regimen will allow for later exposure to the therapeutic vector if needed and block any immuno-toxicity in the CNS. The goal of this study is to measure the safety and efficacy of AAV-mediated gene therapy as a treatment approach for neuronal pathology in Canavan disease. The subject will act as their own control and change from baseline will be assessed in regards to levels of brain NAA, brain water content and morphology, improved clinical status and peripheral levels of NAA. Safety parameters measured in this study will include: serum chemistries and hematology, urinalysis, physical assessments, whole blood assay for vector genomes, immunologic response to ASPA and AAV, as well as reported subject symptom history.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-24 months of age at time of study enrollment
* Have a diagnosis of Canavan disease, as defined by biochemical criteria AND/OR genetic mutation analysis, AND demonstrate clinical findings such as macrocephaly, developmental delay, seizures or other positive findings
* Elevated brain NAA levels, which is correlated with NAA acidemia and aciduria
* Willing to discontinue aspirin, aspirin-containing products and other drugs that may alter platelet function 7 days prior to dosing, resuming 24 hours after the gene transfer agent has been administered

Exclusion Criteria:

* Have required acute (as distinguished from long-term, maintenance or chronic suppressive) oral or intravenous antibiotic therapy for a respiratory infection within 15 days prior to screening
* Have required oral or systemic corticosteroids within the last 15 days prior to baseline screening
* Have a platelet count less than 75,000/mm3
* Have history of platelet dysfunction, evidence of abnormal platelet function at screening, or history of recent use of drugs that may alter platelet function, which the subject is unable/unwilling to discontinue for study agent administration
* Have an INR greater than 1.3
* Have transaminases and alkaline phosphatase more than ten times the upper limit of normal at screening or Day-1; or an abnormal chemistry profile
* Have bilirubin and gamma-glutamyl transpeptidase greater than 2 times the upper limit of normal at screening or Day -1
* Be currently or within the past 30 days participating in any other research protocol involving investigational agents or therapies (Other than approved therapy)
* Have received gene transfer agents within the past 6 months
* Have any other concurrent condition that, in the opinion of the investigator, would make the subject unsuitable for the study.

Ages: 18 Months to 24 Months | Sex: Male
Age Groups: Child
Gender Based: Yes — This is a single patient IND, the patient was previously identified.

CONTACTS AND LOCATIONS:
Overall Officials: Barry J Byrne, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States